CLINICAL TRIAL: NCT05393284
Title: Phase 2 Spectra Study to Evaluate the Safety and Efficacy of OPL-0401 in Patients With Diabetic Retinopathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Valo Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPL-0401-201
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Non-proliferative Diabetic Retinopathy; Proliferative Diabetic Retinopathy
Keywords: diabetic retinopathy; diabetic macular edema; Non-proliferative Diabetic Retinopathy; Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-masked, placebo-controlled, multicenter study to investigate the efficacy and safety of OPL-0401 in patients with diabetes mellitus (DM) with non-proliferative diabetic retinopathy (NPDR) or mild PDR with or without diabetic macular edema (DME). Data from an interim analysis may be used to consider additional arms in the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-masked study in which participants, care providers, central reading center and investigators are masked to study intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OPL-0401 Dose 1 (Experimental): Participants are randomized to OPL-0401 Dose 1 twice daily for 24 weeks
  Interventions: Drug: OPL-0401 Dose 1
- Placebo (Placebo Comparator): Participants are randomized to matching Placebo twice daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPL-0401 Dose 1 — Pharmaceutical Form: Capsule; Route of Administration: Oral
  Arms: OPL-0401 Dose 1
Drug: Placebo — Pharmaceutical Form: Capsule; Route of Administration: Oral
  Arms: Placebo

SUMMARY:
OPL-0401-201 is a multicenter study to investigate the safety and efficacy of OPL-0401 in patients with diabetes mellitus (DM) with diabetic retinopathy.

DETAILED DESCRIPTION:
OPL-0401-201 is a randomized, double-masked, placebo-controlled, multicenter study to investigate the efficacy and safety of OPL-0401 in patients with diabetes mellitus (DM) with NPDR or mild PDR with or without diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria

* Adults ≥ 18 years;
* Diabetes mellitus (type 1, type 2 or other forms);
* Females who are not a woman of childbearing potential (WOCBP) or who agree to use contraception;
* At least one eye with moderately severe to severe NPDR (DRSS levels 47 or 53) or mild PDR (DRSS level 61);
* Patients with or without diabetic macular edema (DME) may be eligible if they meet protocol specified eligibility criteria;
* Best corrected visual acuity (BCVA) early treatment of diabetes retinopathy study (ETDRS) letter score in the study at screening ≥69 letters (approximate Snellen equivalent of 20/40 or better) without CI-DME, or ≥75 letters when CI-DME is present (approximate Snellen equivalent 20/32 or better);
* Anti-vascular endothelial growth factor (VEGF) or any laser treatment is not required nor anticipated in the study eye for least 6 months.

Exclusion Criteria:

* Body mass index ≥ 45 kg/m2
* Uncontrolled diabetes mellitus such as hemoglobin A1c (HbA1C) > 11% or patients who are not currently treated for their diabetes;
* Uncontrolled hypertension defined as systolic > 160mmHg or diastolic > 100 mmHg (despite hypertensive medication);
* Proliferative Diabetes Retinopathy (PDR) with the exception of mild PDR (DRSS 61);
* Evidence of retinal neovascularization (with the exception of mild PDR);
* Any previous Diabetic Retinopathy treatment with focal or grid laser photocoagulation or Pan-Retinal Photocoagulation (PRP);
* History of previously treated DME with fluocinolone acetonide implant (Iluvien®) injection;
* Visual acuity loss due to an ocular condition that would not improve from treatment of DR or resolution of DME (i.e., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, nonretinal condition);
* History of vitreoretinal surgery;
* Intraocular surgery in the study eye within 3 months of randomization or anticipated over the course of the study;
* Uncontrolled glaucoma (e.g. visual field loss or defined as (IOP) ≥ 25 mmHg despite treatment with anti-glaucoma medication);
* Evidence of active infectious blepharitis, keratitis, scleritis, or conjunctivitis in either eye /any intraocular inflammation or infection in either eye within 3 months prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Improvement in Diabetic Retinopathy Severity Scale (DRSS) score | 24 weeks/168 days
  Proportion of patients with a ≥2-step improvement from baseline in DRSS

SECONDARY OUTCOMES:
Proportion of patients with an improvement or worsening in DRSS | 12 Weeks/84 days and 24 Weeks/168 days
  Proportion of patients with an improvement or worsening from baseline in DRSS of ≥ 1, ≥ 2 and ≥ 3 steps
Safety and tolerability | 198 days
  Incidence of Adverse event (AE) and serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Shi, M.D., Study Director — Valo Health, Inc.
Locations (25):
- United States (25):
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants of Southern California, Riverside, California
  - Southern California Permanente Medical Group, Riverside, California
  - Retinal Consultants Medical Group, Sacramento, California
  - California Retina Consultants, Santa Barbara, California
  - Panorama Eye Care, LLC, Fort Collins, Colorado
  - Mid Florida Eye Center, Mt. Dora, Florida
  - Eye Associates of Northeast Louisiana, West Monroe, Louisiana
  - The Retina Care Center, Baltimore, Maryland
  - Massachussetts Eye and Ear, Boston, Massachusetts
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Texas Retina Associates, Dallas, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Austin Retina Associates - Round Rock, Round Rock, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group LLC, Willow Park, Texas
  - Retina Associates of Utah, Salt Lake City, Utah
  - Pacific Northwest Retina, Seattle, Washington
  - Spokane Eye Clinical Research, Spokane, Washington